CLINICAL TRIAL: NCT03671512
Title: A Phase III, Prospective, Randomized, Active Comparator-controlled, Parallel Group, Subject-paired Study Comparing Standard Root Planing vs. a Periodontal Structure Repair Device for Treatment of Pockets Caused by Periodontal Disease.
Brief Title: Standard Root Planing vs. Periodontal Structure Repair Device for Treatment of Pockets Caused by Periodontal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Periovance, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSR-001
Record Dates: First submitted 2018-09-11; First posted 2018-09-14 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: For each subject, one quadrant will be randomized to PSR and the other quadrant will be randomized to conventional scaling and root planing.
Who Masked: Outcomes Assessor
Masking Description: The assessments of efficacy measurements of pocket depth and attachment gain CAL will be performed by a dental professional staff member at the investigator site who is blinded to which procedure was performed in each quadrant. Whenever possible, the same staff member will make these assessments throughout the study. The pocket depth assessments will be performed by a dental professional who has been trained on the actual method. Personnel will be trained to use the University of North Carolina (UNC) probe by the central trainer provided by the sponsor or CRO.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Periodontal Structure Repair (PSR) (Experimental): Periodontal pockets treated with PSR
  Interventions: Device: Periodontal Structure Repair (PSR)
- Standard Root Planing (SRP) (Active Comparator): Periodontal pockets treated with SRP
  Interventions: Device: Standard Root Planing

INTERVENTIONS:
Device: Periodontal Structure Repair (PSR) — Following local anesthesia, initial pocket preparation will be done by bur abrasion utilizing specially designed burs to plane the root surface and remove the inner lining of the pocket. Following bur abrasion, thin strips of gauze sponge are placed into the created space. After removing the gauze strips, PSR is inserted to fill the spaces beginning at the pocket bottom. The final step is placing a layer of cyanoacrylate on both the gingival margin and tooth supragingivally.
  Arms: Periodontal Structure Repair (PSR)
Device: Standard Root Planing — Ultrasonics and hand instruments are used to remove any subgingival deposits on the roots. Standard instruments and standard application are used. Visual or instrument tactile inspection is used to verify the roots are hard-smooth and have been adequately cleaned.
  Arms: Standard Root Planing (SRP)

SUMMARY:
This study evaluates the efficacy and safety of Periodontal Structure Repair device (PSR) compared to conventional periodontal therapy (scaling and root planing) for the treatment of periodontal pockets caused by periodontal disease.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, open, active comparator-controlled study with a parallel group, subject-paired design (i.e. the effect of both treatments can be observed in the same subject).

Subjects must have two quadrants of their mouth that each have at least two teeth with one or more pockets per tooth that are 5-8 mm in depth. Subjects having more than 2 quadrants will have the first 2 quadrants randomized to receive two different treatments (one quadrant root planing and one quadrant PSR procedure) from the group of available quadrants.

Investigators will assess the efficacy of the Periodontal Structure Repair device (PSR) as measured by a reduction in pocket depth.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be in stable health as determined by lack of clinically significant abnormalities as assessed at screening.
2. Subjects must have a minimum of 2 teeth with a pocket depth of 5 to 8 mm per quadrant in at least two quadrants of the mouth with bleeding on probing.
3. Signed and dated informed consent form, meeting all criteria of current FDA regulations and approved by the assigned IRB.
4. Subject must be willing and able to follow all the post treatment oral hygiene requirements.
5. Subjects must be in stable systemic health.

Exclusion Criteria:

1. History of allergy or sensitivity to any of the PSR paste ingredients or other products used in the PSR or Root Planing procedure.
2. Subjects who demonstrate during the pre-treatment prophylaxis cleaning visit that they cannot adequately comply with post treatment dental hygiene requirements of the study.
3. History or current evidence of chronic infectious disease, system disorders, organ dysfunction, cardiovascular disorders, stroke, renal or hepatic disorder, diabetes or bleeding disorders that may prevent the subject from tolerating the scaling and root planing or PSR device and procedure or any significant clinical illness within 90 days of the study start. If any doubt is present regarding the accuracy of the subject's medical history or their suitability to participate, appropriate consultation, e.g., the Chief Medical Officer of InClinca (the CRO) should be sought or the subject excluded.
4. Wears braces or had any dental procedures within 2 weeks of entering the study. Any significant dental issues noted during the screening oral examination. Any ongoing clinically significant trauma or infectious diseases in the oral cavity.
5. Any previous periodontal procedures including scaling and root planing within 6 months of entering the study.
6. Presence of a medical condition requiring regular treatment with antibiotics or treatment with antibiotics within six months prior to entry into the study.
7. Presence of a medical condition requiring treatment with anticoagulant therapy or drugs, such as heparin or warfarin. Subjects prescribed ≤ 325 mg/day of aspirin should not be excluded and this treatment should not be stopped during their participation in this trial.
8. History of psychiatric disorders occurring within the last two years that required hospitalization or medication.
9. Receipt of an Investigational drug as part of a research study within 30 days or 10 half-lives (whichever is longer) prior to entry into the trial.
10. A clinically significant abnormality is detected in the subject's screening blood or urine samples (clinical chemistry, hematology, or urinalysis) that in the opinion of the investigator should prohibit inclusion into the trial.
11. Positive test results for HIV, Hepatitis B surface antigen, or Hepatitis C antibody at screening.
12. Subject is not able to communicate well with the Investigator, to understand and comply with the requirements of the study, or to understand the written informed consent
13. Subject is not suitable to participate in the study in the opinion of the Investigator
14. Teeth with any furcation defects or mobility >2 will be excluded from treatment in both arms of the study.
15. Medication that alters or affects healing such as chemotherapy, immune-suppressive medications within two months of study start.
16. Subjects having received doses of corticosteroids in excess of 20mg per day within 2 months of study start.
17. Subjects who are pregnant or planning to become pregnant during the course/duration of the clinical trial period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Change in periodontal pocket depth compared to standard root planing at 8 weeks | 8 weeks
  The pocket depth is measured using a Williams' periodontal probe. The probe is inserted into the pocket until resistance is met. The depth of the pocket is measured in millimeters (mm) indicated on the probe. Measure the distance from the gingival margin to the tip of the periodontal probe. Each pocket will have six measurement taken around the tooth. The pocket depth measurements to be performed: buccal mesial, buccal, buccal distal, lingual mesial, lingual, lingual distal.
An acceptable safety profile at Visit Week 8 as evidenced by no clinically significant increase in the occurrence of select adverse events | 8 weeks
  The primary safety endpoints are to demonstrate an acceptable safety profile at Visit Week 8 as evidenced by no clinically significant increase in the occurrence of any of the following adverse events for the PSR-treated pockets versus the current standard of treatment for periodontal pockets (scaling and root planing):
  1. an increase in pocket depth ≥ 2 mm
  2. clinical signs and symptoms of an abscess
  3. pain localized to the treated teeth.

SECONDARY OUTCOMES:
Change in periodontal pocket depth compared to standard root planing at 12 and 16 weeks | 12 weeks and 16 weeks
  The pocket depth is measured using a Williams' periodontal probe. Each pocket will have six measurements taken around the tooth at the following locations: buccal mesial, buccal, buccal distal, lingual mesial, lingual, lingual distal.
Change in clinical attachment level compared to standard root planing at Visit Weeks 4, 8, 12 and 16 | 4, 8, 12, 16 weeks
  The gingival margin level measurements to be performed: buccal mesial, buccal, buccal distal, lingual mesial, lingual, lingual distal.
To evaluate the percentage of subjects who achieve 15% and 25% improvements over baseline for pocket depth reduction for PSR-treated versus root-planed teeth. | 4, 8, 12, 16 weeks
  Each pocket will have six measurement taken around the tooth. The pocket depth measurements to be performed include: buccal mesial, buccal, buccal distal, lingual mesial, lingual, lingual distal
To evaluate the percentage of subjects who achieve 15% and 25% improvements over baseline for clinical attachment level for PSR-treated versus root-planed teeth | 4, 8, 12, 16 weeks
  The gingival margin level measurements to be performed: buccal mesial, buccal, buccal distal, lingual mesial, lingual, lingual distal.
Degree of inflammation following procedure | 8 weeks
  Inflammation measured the Gingival Index (Löe and Silness, 1963).
  * 0 = Normal gingiva
  * 1 = Mild inflammation: slight change in color, slight edema. No bleeding on probing.
  * 2 = Moderate inflammation: redness, edema, and glazing. Bleeding on probing.
  * 3 = Severe inflammation: marked redness and edema. Ulceration. Tendency for spontaneous bleeding.
Degree of erythema following procedure | 8 weeks
  Gingival erythema - measured using the Modified Gingival Index (MGI) (Lobene et al. 1986)
  * 0 = absence of inflammation;
  * 1 = mild inflammation or with slight changes in color and texture but not in all portions of gingival marginal or papillary;
  * 2 = mild inflammation, such as the preceding criteria, in all portions of gingival marginal or papillary;
  * 3 = moderate, bright surface inflammation, erythema, edema and/or hypertrophy of gingival marginal or papillary;
  * 4 = severe inflammation: erythema, edema and/or marginal gingival hypertrophy of the unit or spontaneous bleeding, papillary, congestion or ulceration.
Presence or absence of bleeding on probing following procedure | 8 weeks
  Bleeding on probing will be reported by a yes/no response
Degree of Pain using the Pain Quality Assessment Scale (PQAS), National Initiative on Pain Control™ (NIPC). | 8 weeks
  The scoring system will be used to grade the amount of pain felt by the subject in their mouth and jaw areas where the scaling and root planing or PSR treatment was performed.
Gingival Infection: Presence of gingival infection | 8 weeks
  Presence of gingival infection will be recorded by a yes/no response in the case report form. If infection is present, the quadrant of the mouth will be recorded.
Sensitivity | 8 weeks
  Subjects will be asked by the examining dental professional if they have experienced any temperature-related pain or discomfort in their teeth or gums.
Tooth mobility of PSR-treated teeth versus standard root planing | 8 weeks
  Tooth mobility will be assessed using the Tooth Mobility Scale (Miller, 1985)
  * Class 1: <1mm (horizontal) movement of the tooth
  * Class 2: >1mm (horizontal) movement of the tooth
  * Class 3: >1mm (horizontal and vertical mobility) of the tooth
Safety profile of the PSR procedure versus standard root planing for management of periodontal pocket disease through Visit Week 16. | 16 weeks
  The full safety profile will be assessed by the following:
  1. Evaluate the adverse event (AE) safety profile of the PSR procedure versus STA for the management of periodontal pocket disease through the trial.
  2. Evaluate blood laboratory values at Baseline, Visit Week 12 and Visit Week 16.
  3. To evaluate the pocket depth effect of the PSR device and procedure versus STA over time (including 8 week, 12 week and 16 week assessments) utilizing a longitudinal analysis approach.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fare, Study Chair — Periovance, Inc
Locations (4):
- United States (4):
  - University of Alabama at Birmingham School of Dentistry, Birmingham, Alabama
  - Forsyth Institute, Cambridge, Massachusetts
  - Stony Brook School of Dental Medicine, Stony Brook, New York
  - University of North Carolina at Chapel Hill School of Dentistry, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No